CLINICAL TRIAL: NCT02517268
Title: A Prospective Randomized Controlled Trial Evaluating an Accelerated 5 Day Pathway for Discharge Following Pancreaticoduodenectomy (PD): Whipple Accelerated Recovery Pathway (WARP Trial)
Brief Title: Accelerated Recovery Pathway for Discharge After Surgery in Patients With Pancreatic Cancer
Acronym: WARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15D.050; 2014-082 (Other: CCRRC); JT 6901 (Other: JeffTrial Number)
Record Dates: First submitted 2015-07-30; First posted 2015-08-06 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard 7-Day Pathway (Active Comparator): Patients follow the standard 7-day pathway following pancreaticoduodenectomy
  Interventions: Procedure: Pancreaticoduodenectomy
- Accelerated 5-Day Pathway (Experimental): Patients follow the Whipple accelerated 5-day pathway following pancreaticoduodenectomy. The accelerated pathway includes more rapidly leaving the ICU setting, early mobilization and enhanced physical therapy, multimodal pain control, dietary modifications, and increased and standardized phone contact by a nurse practitioner during the first week following hospital discharge.
  Interventions: Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy
  Other Names: Pancreatoduodenectomy; Whipple procedure; Kausch-Whipple procedure

SUMMARY:
This randomized clinical trial studies accelerated recovery pathway for discharge after surgery in patients with pancreatic cancer. A standardized accelerated recovery pathway may improve outcomes after surgery following complex abdominal operations resulting in a shorter length of stay in patients with pancreatic cancer. It may also help patients to mobilize more quickly and return to the home setting, decrease hospital-acquired infectious complications, and increase potential cost savings. It is not yet known whether an accelerated recovery pathway is better than a standard recovery pathway for discharge following surgery in patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The use of an accelerated pathway will result in a shorter postoperative hospital length of stay for patients undergoing pancreaticoduodenectomy (PD) without an increase in perioperative complications or readmission rates.

SECONDARY OBJECTIVES:

I. The investigators anticipate lower cost, lower readmission rate, similar rate of post-operative complications (delayed gastric emptying [DGE], anastomotic leaks, intra-abdominal abscesses, wound infection, urinary tract infection [UTI], respiratory compromise, renal failure, etc.) in our study group.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients follow the standard 7-day pathway at the end of surgery.

ARM II: Patients follow the Whipple accelerated 5-day pathway at the end of surgery. The accelerated pathway includes more rapidly leaving the ICU setting, early mobilization and enhanced physical therapy, multimodal pain control, dietary modifications, and increased and standardized phone contact by a nurse practitioner during the first week following hospital discharge.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Pancreaticoduodenectomy
2. Firm gland texture
3. Subjects able to provide informed consent

Exclusion Criteria:

1. Preoperative factors:

   * Congestive heart failure (CHF)
   * End stage renal disease (ESRD)
   * Chronic obstructive pulmonary disease (COPD)
   * Pregnancy
   * Albumin < 3 gm/dL
   * Poor preoperative performance status as defined by: timed get up and go (< 15 seconds)
   * Patients cannot be homeless or have substance dependence
2. Intraoperative factors:

   * Estimated blood loss (EBL) > 1 liter
   * Failure to extubate at the conclusion of the case
   * Operative time > 8 hours
   * Need for vascular resection/reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harish Lavu, MD, Study Chair — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lavu H, McCall NS, Winter JM, Burkhart RA, Pucci M, Leiby BE, Yeo TP, Cannaday S, Yeo CJ. Enhancing Patient Outcomes while Containing Costs after Complex Abdominal Operation: A Randomized Controlled Trial of the Whipple Accelerated Recovery Pathway. J Am Coll Surg. 2019 Apr;228(4):415-424. doi: 10.1016/j.jamcollsurg.2018.12.032. Epub 2019 Jan 17. PMID 30660818
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 participants were not included in the final analysis as they were not randomized to either arm of the study. Prior to randomization, 3 participants withdrew consent, and 19 participants did not undergo their procedure at Thomas Jefferson University Hospital
Pre-assignment Details: 22 participants were not included in the final analysis as they were not randomized to either arm of the study. Prior to randomization, 3 participants withdrew consent, and 19 participants did not undergo their procedure at Thomas Jefferson University Hospital. On the control arm, 1 participant withdrew consent after randomization
Groups:
- Standard 7-Day Pathway: Patients follow the standard 7-day pathway following pancreaticoduodenectomy
  Pancreaticoduodenectomy
- Accelerated 5-Day Pathway: Patients follow the Whipple accelerated 5-day pathway following pancreaticoduodenectomy. The accelerated pathway includes more rapidly leaving the ICU setting, early mobilization and enhanced physical therapy, multimodal pain control, dietary modifications, and increased and standardized phone contact by a nurse practitioner during the first week following hospital discharge.
  Pancreaticoduodenectomy
Period: Overall Study
Arm/Group | Standard 7-Day Pathway | Accelerated 5-Day Pathway
Started | 40 | 37
Completed | 39 | 37
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard 7-Day Pathway | Accelerated 5-Day Pathway | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 15 | 33
  >=65 years | 21 | 22 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 17 | 20 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 36 | 35 | 71
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 34 | 36 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Discharged by Post-operative Day 5
Description: Two-sided alpha 0.05 will be used to detect a increase in the percentage of patients discharged on post-operative day 5
Time Frame: Up to post-operative day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Standard 7-Day Pathway | Accelerated 5-Day Pathway
Number analyzed (Participants) | 39 | 37
Participants | 5 | 28

2. Secondary Outcome: Post-operative Median Length of Stay
Time Frame: 30 days after operation
Measure: Median (Full Range); unit: days
Arm/Group | Standard 7-Day Pathway | Accelerated 5-Day Pathway
Number analyzed (Participants) | 39 | 37
days | 6 [5 to 23] | 5 [4 to 11]

3. Secondary Outcome: Cost
Description: Cost will be assessed by reviewing inpatient hospital charges
Time Frame: 30 days after operation
Measure: Median (Full Range); unit: US Dollar
Arm/Group | Standard 7-Day Pathway | Accelerated 5-Day Pathway
Number analyzed (Participants) | 39 | 37
US Dollar | 155,542 [125,519 to 398,764] | 139,735 [104,689 to 253,830]

4. Secondary Outcome: Readmission Rate
Time Frame: 30 days after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard 7-Day Pathway | Accelerated 5-Day Pathway
Number analyzed (Participants) | 39 | 37
Participants | 4 | 3

5. Secondary Outcome: Incidence of Post-operative Complications (DGE, Anastomotic Leaks, Intra-abdominal Abscesses, Wound Infection, UTI, Respiratory Compromise, Renal Failure, Etc.)
Time Frame: 30 days after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard 7-Day Pathway | Accelerated 5-Day Pathway
Number analyzed (Participants) | 39 | 37
Participants
  Delayed Gastric Emptying (DGE) | 13 | 5
  Anastomotic leaks | 0 | 0
  intra-abdominal abscess | 1 | 1
  Wound Infection | 1 | 0
  Urinary Tract Infection (UTI) | 2 | 1
  Pancreatic Fistula | 2 | 4
  Renal Failure | 0 | 0
  Cardiovascular | 0 | 1
  Pulmonary | 3 | 0
  Deep Vein Thrombosis | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline to 3 months after surgery
Arm/Group | Standard 7-Day Pathway | Accelerated 5-Day Pathway
All-Cause Mortality (participants affected / at risk) | 10/39 | 13/37
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/37
Other Adverse Events (participants affected / at risk) | 17/39 | 5/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard 7-Day Pathway (N=39) | Accelerated 5-Day Pathway (N=37)
Delayed Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard 7-Day Pathway (N=39) | Accelerated 5-Day Pathway (N=37)
Pancreatic Fistula (Gastrointestinal disorders) | 3 | 1
Delayed Gastric Emptying (Gastrointestinal disorders) | 9 | 3
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT02517268/Prot_SAP_000.pdf